CLINICAL TRIAL: NCT05256654
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of LY3561774 in Adults With Mixed Dyslipidemia
Brief Title: A Study of LY3561774 in Participants With Mixed Dyslipidemia
Acronym: PROLONG-ANG3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18361; J3F-MC-EZCB (Other: Eli Lilly and Company); 2021-005407-13 (EudraCT Number)
Record Dates: First submitted 2022-02-23; First posted 2022-02-25 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases; Hyperlipoproteinemia
Keywords: Triglycerides; LDL Cholesterol; Mixed Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases; Hyperlipoproteinemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3561774 100 mg (Experimental): Participants received 100 milligram (mg) LY3561774 subcutaneously (SC) on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
  Interventions: Drug: LY3561774
- LY3561774 400 mg (Experimental): Participants received 400 mg LY3561774 SC on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
  Interventions: Drug: LY3561774
- LY3561774 800 mg (Experimental): Participants received 800 mg LY3561774 SC on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
  Interventions: Drug: LY3561774
- Placebo (Placebo Comparator): Participants received placebo SC on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3561774 — Administered SC
  Other Names: Solbinsiran
  Arms: LY3561774 100 mg; LY3561774 400 mg; LY3561774 800 mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This a multicenter, Phase 2b, double-blind, placebo-controlled, parallel group study to provide data on efficacy and safety of LY3561774 administered subcutaneously at various doses in participants with mixed dyslipidemia and on a stable dose of a statin.

ELIGIBILITY:
Inclusion Criteria:

* Have fasting triglycerides (TGs) within the range of 150 (1.69 millimole/liter (mmoL) to 499 milligram/deciliter (mg/dL) 2.26 to 5.64 millimole/liter (mmol/L) at screening.
* Have fasting LDL-C ≥70 mg/dL (1.81 mmol/L) at screening.
* Have non-HDL-C ≥ 130 mg/dL (3.36 mmol/L) at screening.
* Must be on a stable moderate or high-intensity dose of a statin for at least 2 months before screening and remain on the same medication and dose for the duration of the study.
* Have a body mass index within the range of 18.5 to 40.0 kilogram/square meter (kg/m²), inclusive

Exclusion Criteria:

* Have in the 6 months prior to screening, uncontrolled Type 1 or Type 2 diabetes, defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization, or have an hemoglobin A1c (HbA1c) ≥8% at screening.
* Have a history of nephrotic syndrome.
* Have a history of acute or chronic pancreatitis.
* Have had within the past 3 months prior to screening

  * Myocardial infarction
  * Unstable angina
  * Coronary artery bypass graft
  * Percutaneous coronary intervention - diagnostic angiograms are permitted
  * Peripheral artery disease
  * Transient ischemic attack, or
  * Cerebrovascular accident
* Have New York Heart Association Class III or IV heart failure or last known left ventricular ejection fraction <30%.
* Have undergone LDL apheresis within 12 months prior to screening.
* Have clinically relevant anemia, as defined by the investigator.
* Have, within 1 year prior to screening or plan on having during the study, surgical treatment for obesity.
* Have within 3 years prior to screening a history of chronic alcohol abuse, IV drug abuse, or other illicit drug abuse.
* Have uncontrolled hypertension.
* Have used or are taking products for the purpose of lowering lipid levels (except for statins, PCSK9 inhibitors, bempedoic acid, and ezetimibe). This includes lipid-regulating medication, over-the-counter products, or herbal therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (41):
- United States (6):
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - MD Medical Research, Oxon Hill, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Premier Research, Trenton, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
- Argentina (10):
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Air
  - Glenny Corp, Buenos Aires, Ciudad Aut
  - CIPREC, CABA, Ciudad Aut
  - Investigaciones Medicas Imoba Srl, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Ciudad Autónoma de Buenos Aire
  - Sanatorio San Martin, Venado Tuerto, Santa Fe Province
  - Fundación Respirar, Buenos Aires
  - Clínica Privada Velez Sarsfield, Córdoba
  - Centro de Investigaciones Clinicas Instituto del Corazon (CICIC), Córdoba
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Canada (5):
  - OCT Research ULC, Kelowna, British Columbia
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Viacar Recherche Clinique, Greenfield Park, Quebec
  - Clinique des Maladies Lipidiques de Québec, Québec, Quebec
- Japan (4):
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Heishinkai Medical Group ToCROM Clinic, Shinjuku-ku, Tokyo
  - AMC Nishiumeda Clinic, Osaka
- Mexico (5):
  - Virgen Cardiovascular Research SC, Guadalajara, Jalisco
  - Cardiolink Clin Trials, Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
- Poland (5):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz, Kujawsko-p
  - Niepubliczny Zakład Opieki Zdrowotnej "Przychodnia z Sercem", Grojec, Lesser Poland Voivodeship
  - Centrum Zdrowia Tuchów, Wierzchosławice, Lesser Poland Voivodeship
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
- Turkey (Türkiye) (6):
  - Ege Universitesi Hastanesi, Bornova, İzmir
  - Necmettin Erbakan Meram Medical Fac., Meram, Konya
  - Akdeniz Universitesi Hastanesi, Antalya
  - Istanbul University Cerrahpasa Medical School Internal Diseases Institute, Istanbul
  - Kocaeli Üniversitesi, Kocaeli
  - Mersin University, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Ray KK, Oru E, Rosenson RS, Jones J, Ma X, Walgren J, Haupt A, Verma S, Gaudet D, Nicholls SJ, Ruotolo G. Durability and efficacy of solbinsiran, a GalNAc-conjugated siRNA targeting ANGPTL3, in adults with mixed dyslipidaemia (PROLONG-ANG3): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet. 2025 May 3;405(10489):1594-1607. doi: 10.1016/S0140-6736(25)00507-0. Epub 2025 Mar 31. PMID 40179932
- See also: A Study of LY3561774 in Participants With Mixed Dyslipidemia (PROLONG-ANG3) — https://trials.lillytrialguide.com/en-US/trial/1g8CjEO0knBk2QA03EkpaY

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo subcutaneously (SC) on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
- LY3561774 100 mg: Participants received 100 mg LY3561774 SC on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
Period: Overall Study
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Started | 58 | 30 | 58 | 59
Received at Least 1 Dose of Study Drug | 57 | 30 | 58 | 59
Completed | 57 | 27 | 55 | 54
Not Completed | 1 | 3 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 3
Not completed — Earthquake at the Turkey site prevented participation in the study | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg | Total
Number analyzed (Participants) | 58 | 30 | 58 | 59 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.50 (11.61) | 58.40 (10.97) | 56.40 (11.97) | 57.30 (10.61) | 56.70 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 18 | 29 | 29 | 111
  Male | 23 | 12 | 29 | 30 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 20 | 39 | 44 | 139
  Not Hispanic or Latino | 22 | 8 | 19 | 15 | 64
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 21 | 11 | 14 | 22 | 68
  Asian | 11 | 6 | 10 | 9 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 25 | 13 | 34 | 28 | 100
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 15 | 8 | 21 | 18 | 62
  Canada | 5 | 4 | 7 | 2 | 18
  Japan | 7 | 4 | 7 | 7 | 25
  Mexico | 21 | 12 | 18 | 26 | 77
  Poland | 3 | 0 | 1 | 1 | 5
  Turkey | 3 | 2 | 3 | 3 | 11
  United States | 4 | 0 | 1 | 2 | 7
Baseline Apolipoprotein B (ApoB) [Median (Full Range); unit: milligram per deciliter (mg/dL)] — Population: Number of participants with non-missing data, used as denominator
  milligram per deciliter (mg/dL)
    number analyzed (Participants) | 56 | 30 | 58 | 59 | 203
    (all) | 111 [23 to 246] | 109.50 [49 to 186] | 112 [73 to 169] | 114 [52 to 205] | 111 [23 to 246]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline for Apolipoprotein B (ApoB) at Day 180
Description: Change in apoB levels from baseline to Day 180 expressed as a percentage of the baseline levels. Least Square Mean (LS mean) using Mixed Model for Repeated Measures (MMRM) model adjusted for baseline.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable apoB values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -11.6 (3.65) | -14.1 (4.98) | -24.3 (3.10) | -19.0 (3.35)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.691, Mixed Models Analysis; Mean Difference (Net) = -2.8, 95% CI 2-sided [-15.5 to 11.9], Standard Error of Mean 6.92 — Model uses log-transformed outcome and baseline variables, including terms for baseline, strata (Triglycerides (TG) <250 milligram per deciliter (mg/dL) or >=250 mg/dL at screening), and the interaction between treatment and time
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -14.3, 95% CI 2-sided [-23.6 to -3.9], Standard Error of Mean 4.98 — Model uses log-transformed outcome and baseline variables, including terms for baseline, strata (TG <250 mg/dL or >=250 mg/dL at screening), and the interaction between treatment and time
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p = 0.140, Mixed Models Analysis; Mean Difference (Net) = -8.3, 95% CI 2-sided [-18.3 to 2.9], Standard Error of Mean 5.36 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percent Change From Baseline for Angiopoietin-like Protein 3 (ANGPTL3) at Day 180
Description: Change in ANGPTL3 levels from baseline to Day 180 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable ANGPTL3 values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -3.2 (6.22) | -55.7 (4.01) | -70.8 (1.86) | -77.3 (1.46)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -54.3, 95% CI 2-sided [-63.3 to -43.1], Standard Error of Mean 5.08 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -69.8, 95% CI 2-sided [-74.8 to -63.9], Standard Error of Mean 2.73 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -76.6, 95% CI 2-sided [-80.4 to -72.0], Standard Error of Mean 2.13 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percent Change From Baseline for Low Density Lipoprotein-Cholesterol (LDL-C) at Day 180
Description: Change in LDL-C levels from baseline to the day 180 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable LDL-C direct values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -8.7 (3.87) | -9.9 (5.39) | -24.0 (3.21) | -19.7 (3.42)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.854, Mixed Models Analysis; Mean Difference (Net) = -1.3, 95% CI 2-sided [-14.6 to 14.0], Standard Error of Mean 7.24 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p = 0.002, Mixed Models Analysis; Mean Difference (Net) = -16.8, 95% CI 2-sided [-26.0 to -6.4], Standard Error of Mean 4.98 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Net) = -12.1, 95% CI 2-sided [-21.9 to -1.1], Standard Error of Mean 5.28 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percent Change From Baseline for High Density Lipoprotein-Cholesterol (HDL-C) at Day 180
Description: Change in HDL-C levels from baseline to the Day 180 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable HDL-C values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | 4.3 (2.59) | -2.1 (3.43) | -12.8 (2.15) | -19.4 (2.00)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.143, Mixed Models Analysis; Mean Difference (Net) = -6.1, 95% CI 2-sided [-13.8 to 2.2], Standard Error of Mean 4.03 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -16.4, 95% CI 2-sided [-22.0 to -10.5], Standard Error of Mean 2.93 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -22.7, 95% CI 2-sided [-27.9 to -17.2], Standard Error of Mean 2.71 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Percent Change From Baseline for Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) at Day 180
Description: Change in non-HDL-C levels from baseline to the Day 180 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable Non HDL-C values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- LY3561774 400 mg: Participants received 200 mg LY3561774 SC on Day 0 and Day 90 (-5 to +10 days). Follow up was continued until Day 360.
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -10.2 (3.24) | -19.8 (4.06) | -33.1 (2.41) | -31.5 (2.47)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.068, Mixed Models Analysis; Mean Difference (Net) = -10.8, 95% CI 2-sided [-21.1 to 0.9], Standard Error of Mean 5.55 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -25.5, 95% CI 2-sided [-32.6 to -17.6], Standard Error of Mean 3.79 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -23.8, 95% CI 2-sided [-31.1 to -15.7], Standard Error of Mean 3.88 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percent Change From Baseline for Triglycerides at Day 180
Description: Change in triglycerides levels from baseline to the Day 180 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 180
Population: All randomized participants receiving at least 1 dose of study drug with evaluable triglycerides values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -15.1 (4.01) | -45.9 (3.61) | -57.8 (1.98) | -59.7 (1.90)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -36.3, 95% CI 2-sided [-45.8 to -25.1], Standard Error of Mean 5.21 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -50.3, 95% CI 2-sided [-56.4 to -43.3], Standard Error of Mean 3.31 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -52.5, 95% CI 2-sided [-58.4 to -45.9], Standard Error of Mean 3.17 — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Percent Change From Baseline for Angiopoietin-like Protein 3 (ANGPTL3)
Description: Change in ANGPTL3 levels from baseline to Day 270 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 270
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -17.0 (6.00) | -49.0 (5.28) | -61.9 (2.75) | -69.8 (2.19)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -38.6, 95% CI 2-sided [-52.2 to -21.2], Standard Error of Mean 7.76 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -54.0, 95% CI 2-sided [-62.4 to -43.8], Standard Error of Mean 4.69 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -63.6, 95% CI 2-sided [-70.3 to 55.5], Standard Error of Mean 3.72 — [estimate comment as in outcome 1, analysis 2]

8. Secondary Outcome: Percent Change From Baseline for Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C)
Description: Change in non-HDL-C levels from baseline to the Day 270 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 270
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -9.8 (3.22) | -13.5 (4.44) | -27.6 (2.56) | -27.3 (2.59)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.506, Mixed Models Analysis; Mean Difference (Net) = -4.1, 95% CI 2-sided [-15.2 to 8.5], Standard Error of Mean 5.99 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -19.7, 95% CI 2-sided [-27.2 to -11.3], Standard Error of Mean 4.04 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -19.4, 95% CI 2-sided [-27.0 to -11.0], Standard Error of Mean 4.06 — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Percent Change From Baseline for High Density Lipoprotein-Cholesterol (HDL-C)
Description: Change in HDL-C levels from baseline to the Day 270 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 270
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | 1.5 (2.48) | -1.9 (3.48) | -7.3 (2.24) | -10.9 (2.18)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.428, Mixed Models Analysis; Mean Difference (Net) = -3.4, 95% CI 2-sided [-11.2 to 5.2], Standard Error of Mean 4.16 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p = 0.009, Mixed Models Analysis; Mean Difference (Net) = -8.7, 95% CI 2-sided [-14.7 to -2.3], Standard Error of Mean 3.14 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -12.2, 95% CI 2-sided [-18.0 to -6.0], Standard Error of Mean 3.04 — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Percent Change From Baseline for Low Density Lipoprotein-Cholesterol (LDL-C)
Description: Change in LDL-C levels from baseline to the day 270 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 270
Population: All randomized participants receiving at least 1 dose of study drug with evaluable LDL-C values at baseline, and at least 1 post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -12.7 (3.78) | -7.1 (5.81) | -21.0 (3.39) | -17.5 (3.57)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.412, Mixed Models Analysis; Mean Difference (Net) = 6.5, 95% CI 2-sided [-8.4 to 23.7], Standard Error of Mean 8.10 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p = 0.104, Mixed Models Analysis; Mean Difference (Net) = -9.5, 95% CI 2-sided [-19.7 to 2.1], Standard Error of Mean 5.52 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p = 0.363, Mixed Models Analysis; Mean Difference (Net) = -5.4, 95% CI 2-sided [-16.2 to 6.7], Standard Error of Mean 5.79 — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Percent Change From Baseline for Apolipoprotein B (ApoB)
Description: Change in apoB levels from baseline to Day 270 expressed as a percentage of the baseline levels. LS mean using MMRM model adjusted for baseline.
Time Frame: Baseline, Day 270
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -9.5 (3.57) | -19.2 (4.61) | -19.7 (3.18) | -19.4 (3.20)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p = 0.101, Mixed Models Analysis; Mean Difference (Net) = -10.8, 95% CI 2-sided [-22.2 to 2.3], Standard Error of Mean 6.19 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p = 0.033, Mixed Models Analysis; Mean Difference (Net) = -11.3, 95% CI 2-sided [-20.6 to -1.0], Standard Error of Mean 4.96 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p = 0.040, Mixed Models Analysis; Mean Difference (Net) = -10.9, 95% CI 2-sided [-20.3 to -0.6], Standard Error of Mean 4.98 — [estimate comment as in outcome 1, analysis 2]

12. Secondary Outcome: Percent Change From Baseline for Triglycerides
Description: Change in triglycerides levels from baseline to the Day 270 expressed as a percentage of the baseline levels. LS Mean from MMRM model adjusted for baseline and treatment.
Time Frame: Baseline, Day 270
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 57 | 30 | 58 | 59
Percent change | -13.9 (4.63) | -38.3 (4.80) | -50.5 (2.63) | -52.5 (2.55)
Statistical Analysis 1: Comparison: Placebo vs LY3561774 100 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -28.3, 95% CI 2-sided [-40.5 to -13.6], Standard Error of Mean 6.79 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs LY3561774 400 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -42.5, 95% CI 2-sided [-50.5 to -33.2], Standard Error of Mean 4.35 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs LY3561774 800 mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -44.8, 95% CI 2-sided [-52.5 to -35.9], Standard Error of Mean 4.20 — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Pharmacokinetics (PK): Seady State Area Under the Concentration Curve From Hour 0 Extrapolated to Infinity (AUC 0-∞) of LY3561774
Description: PK: Seady State AUC (0-∞) of LY3561774
Time Frame: On Day 0: 0.5 hour (hr) and at the latest time after 2 hr post-dose, Day 90: 24 to 48 hr postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hour per milliliter (ng*h/mL)
Arm/Group | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
Number analyzed (Participants) | 30 | 58 | 59
nanogram.hour per milliliter (ng*h/mL) | 6979 (35) | 25045 (24) | 61306 (43)

ADVERSE EVENTS:
Time Frame: Baseline up to 360 Days
Description: All participants who received at least one dose of the study drug, regardless of their eligibility for the study.
Arm/Group | Placebo | LY3561774 100 mg | LY3561774 400 mg | LY3561774 800 mg
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/30 | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 5/57 | 1/30 | 3/58 | 2/59
Other Adverse Events (participants affected / at risk) | 16/57 | 14/30 | 14/58 | 9/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | LY3561774 100 mg (N=30) | LY3561774 400 mg (N=58) | LY3561774 800 mg (N=59)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=57) | LY3561774 100 mg (N=30) | LY3561774 400 mg (N=58) | LY3561774 800 mg (N=59)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Covid-19 (Infections and infestations) | 4 (4) | 4 (4) | 3 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Pancreatic enzymes increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05256654/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT05256654/SAP_001.pdf